CLINICAL TRIAL: NCT06562491
Title: Phenotypes Associated With Constitutional EGFR Pathogenic Variants
Acronym: EGFRench
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP240782
Record Dates: First submitted 2024-07-19; First posted 2024-08-20 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2024-07

CONDITIONS: Bronchopulmonary Cancers; Constitutional EGFR
Keywords: Phenotypes; constitutional; EGFR

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
A small proportion of lung cancers are hereditary, i.e. caused by a constitutional pathogenic variant (PV). EGFR " Epidermal Growth Factor Receptor " is a major cancer predisposing gene, mainly via the T790M variant. The study aims to collect French national data on EGFR pathogenic variant carriers (affected and unaffected), in order to better characterise the associated phenotypes.

A retrospective, multicenter cohort study will be carried out. The study aims to include 20 to 25 patients identified as EGFR pathogenic variant carriers between 2018 and 2024. Data will be gathered from either paper or electronic patient files from the Oncogenetics clinics or laboratory. Eligible patients will be informed and given a possibility to opt out. Of note, all previously signed a consent form for genetic testing. Each participating centre will be responsible for transcribing the pseudonymised data from its patients' medical records into a secure Excel file unique to each centre. The anonymized data obtained from the patient files will be electronically stored in a secure document accessible only to the principal investigator and a maximum of two close collaborators involved in the study. Data will be sent by participating centres to investigators from the Medical Genetics Department at APHP Sorbonne via the secure national RENATER platform for analysis.

A Simple description of the cohort, e.g. mean/median age, proportion and type of somatic changes, prevalence of smoking will be done.

DETAILED DESCRIPTION:
A small proportion of lung cancers, particularly adenocarcinomas, is hereditary. Hereditary lung cancers occur in individuals with a genetic predisposition to the disease. It is important to remember that a proportion of non-small cell lung cancers develop in never smokers, illustrating the importance of other risk factors, such as pollution, radon or genetic factors. The overall proportion of hereditary lung adenocarcinomas is low, probably around 1%. On a French national scale, this still represents a few hundred cases per year.

EGFR is now an established susceptibility gene. EGFR variants are best known as somatic variants, as markers of sensitivity or resistance to tyrosine kinase inhibitors (TKIs).EGFR T790M, in particular, is usually an acquired variant seen in patients exposed to 1st and 2nd-generation tirosine kinase inihibitors (erlotinib, gefitinib, afatinib). But it is also sometimes constitutional, in which case it is somatically observed at diagnosis, when the patient has not be prescribed a TKI yet. Our research aims to gather data on French EGFR pathogenic variant carriers, i.e, index cases and relatives (affected and unaffected), and to describe the related phenotypes.

A retrospective, multicenter cohort study will be carried out,. The study aims to include 20 to 25 EGFR pathogenic variant carriers identified as such between 2018 and 2024. Data will be gathered from either paper or electronic patient files from the Oncogenetics clinic or laboratory, Eligible patients will be informed and given a possibility to opt out, in conformity with French legal requirements. Of note, all previously signed a consent form for genetic testing. . Each participating centre will be responsible for transcribing the pseudonymised data from its patients' medical records into a secure Excel file unique to each centre. The anonymized data obtained from the patient files will be electronically stored in a secure document accessible only to the principal investigator and a maximum of two close collaborators involved in the study. Data will be sent by participating centres to investigators from the Medical Genetics Department at APHP Sorbonne via the secure national RENATER platform.

Descriptive statistics will be done to describe the cohort's characeristics, e.g. mean/median age, proportion and type of somatic changes, prevalence of smoking in order to better characterize the phenotypes associated with EGFR.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 ans
* Carrier of a constitutional pathogenic variant of the EGFR gene
* Social security beneficiary, excluding AME

Exclusion Criteria:

* Guardianship or curatorship
* Opposition to the use of data

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Carrier of a constitutional pathogenic variant of the EGFR gene
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
average/median, proportion and type of somatic disorders, prevalence of smoking | Through out study 12 months

IPD SHARING:
Plan to Share IPD: Yes
The procedures carried out with the French data privacy authority (CNIL) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.